CLINICAL TRIAL: NCT02080936
Title: Does Muscle Wasting Always Mean Muscle Weakness? A Prevalence Study in COPD
Acronym: M2W
Status: Completed | Type: Observational
Sponsor: 5 Santé (Other)
Responsible Party: Sponsor
Other Study IDs: FVIE_M2W
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: COPD
Keywords: Experimental approaches; Peripheral muscle Keyword; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Peripheral muscle mass and strength are relevant indicators of COPD survival. Current guidelines recommend to assess muscle strength only in muscle wasted patients. However, a recent study reported quadriceps weakness without muscle wasting (Menon, M et al. Resp. Res.2012, 13:119). Thus, these guidelines raise the risk to miss out some weak patients. In clinical settings, fat-free-mass index (FFMI) is indicated as a simple index to assess muscle wasting. We aimed at determining the prevalence of patients entering in pulmonary rehabilitation (PR) a priori not eligible for muscle strength evaluation given the lack of muscle wasting clinical signs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have got FFMI (bioimpedance)
* Patients who have done quadriceps muscle strenght evaluation

Exclusion Criteria:

* Patients without FFMI
* Patients without quadriceps muscle strenght

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COPD patients from "Clinique du Souffle La vallonie" and "Clinique du Souffle La Solane"
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Muscle wasting in COPD patient | baseline

SECONDARY OUTCOMES:
Muscle weakness in COPD patient | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du Souffle La Vallonie, Lodève, France